CLINICAL TRIAL: NCT06697405
Title: Incidence, Risk Factors, and Outcomes of Gastrointestinal Complications in Patients Undergoing Heart Valve Replacement With Cardiopulmonary Bypass
Brief Title: Impact of Cardiopulmonary Bypass Time on Gastrointestinal Complications
Status: Completed | Type: Observational
Sponsor: Hepatopancreatobiliary Surgery Institute of Gansu Province (Other)
Responsible Party: Principal Investigator, Wenbo Meng, Director of Surgery, Hepatopancreatobiliary Surgery Institute of Gansu Province
Other Study IDs: CPB-GICs
Record Dates: First submitted 2024-11-16; First posted 2024-11-20 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Valvular Disease
Keywords: Cardiopulmonary bypass; Gastrointestinal injury; Valvular disease; Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CPB time ≥ 120 minutes: Patients will be grouped into a prolonged CPB group (CPB ≥120 minutes)
  Interventions: Other: Prolonged ≥ 120 minutes
- CPB time < 120 minutes: Patients will be grouped into a normal CPB group (CPB <120 minutes) .
  Interventions: Other: Prolonged ≥ 120 minutes

INTERVENTIONS:
Other: Prolonged ≥ 120 minutes — No intervention, regular therapy

SUMMARY:
This retrospective study investigates the relationship between cardiopulmonary bypass (CPB) duration and the incidence of gastrointestinal complications (GICs) in patients undergoing heart valve replacement. Patients will be grouped into a normal CPB group (CPB <120 minutes) and a prolonged CPB group (CPB ≥120 minutes). The study aims to determine whether prolonged CPB time is associated with a higher risk of GICs and to evaluate the outcomes and recovery process for patients who develop GICs postoperatively.

DETAILED DESCRIPTION:
Heart valve replacement with CPB carries a risk of GICs due to potential ischemia-reperfusion injury to the gastrointestinal tract. GICs in the postoperative period can lead to increased morbidity and prolong recovery. Prolonged CPB time may serve as a predictive factor for the development of GICs following heart valve replacement. This study will utilize established diagnostic criteria to define GICs, which include clinical symptoms, laboratory tests, and imaging as necessary, based on standards from critical care and gastrointestinal surgery guidelines. By understanding this correlation, the study aims to reduce the incidence and severity of postoperative GICs and improve surgical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing heart valve replacement with CPB
* Age ≥ 18 years and ≤ 75 years

Exclusion Criteria:

* Have received major gastrointestinal surgery within 5 years.
* History of severe infection (e.g., pneumonia, urinary tract infection) requiring hospitalization within 1 month prior to surgery.
* Inflammatory bowel disease (IBD), including ulcerative colitis, Crohn's disease, or colitis.
* Acute gastroenteritis.
* Clostridium difficile or Helicobacter pylori infection.
* Chronic constipation.
* Peptic ulcer.
* Polyps in the stomach or intestines.
* Gastrointestinal neoplasms.
* Abdominal hernia.
* Irritable bowel syndrome.
* Acute or chronic cholecystitis, hepatitis.
* Patients who died intraoperatively or within 24 hours postoperatively.
* Patients with digestive system tumors.
* Pregnancy or breastfeeding could affect postoperative medication use and study observations.
* Involvement in other studies that may interfere with the objective results of this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing heart valve replacement with differ CPB durations.
Sampling Method: Non-Probability Sample
Enrollment: 1444 (Actual)
Dates: Start 2024-12-24 (Actual); Primary Completion 2025-12-25 (Actual); Study Completion 2025-12-25 (Actual)

PRIMARY OUTCOMES:
The acute gastrointestinal injury (AGI) score | 1 month
  The AGI score of the patient within the seventh postoperative day was performed daily according to the European Society of critical care (2012) guidelines for AGI. Determined the severity with grade 1-4,The higher the score, the more serious it is.

SECONDARY OUTCOMES:
Return Time of Bowel Sounds | 1 month
  The time to first detection of bowel sounds after surgery, monitored daily in the morning and evening by auscultation.
Frequency of Bowel Sounds | 1 month
  The number of bowel sounds counted at 12-hour intervals, recorded twice daily to assess gastrointestinal motility.
Time to First Defecation | 1 month
  The time to the first defecation was asked morning and evening after surgery.
Proportion of Cocci and Bacilli in Feces | 1 month
  Analysis of bacterial composition in the first stool sample post-surgery, focusing on the ratio of cocci to bacilli.
5.C-Reactive Protein (CRP) | 1 month
  Maximum CRP level recorded within the first week after surgery.
Procalcitonin (PCT) | 1 month
  Maximum PCT level recorded within the first week after surgery.
Alanine Aminotransferase (ALT) | 1 month
  The investigators defined it as the maximum value of ALT within 7 days after surgery.
Aspartate Aminotransferase (AST) | 1 month
  The investigators defined it as the maximum value of ALT within 7 days after surgery.
Creatinine | 1 month
  The investigators defined it as the maximum value of Creatinine within 7 days after surgery.
Left Ventricular Ejection Fraction (LVEF) | 1 month
  LVEF assessed through echocardiography on days 1 and 3 post-surgery to monitor cardiac function.
Ventilator assisted time (VAT) | 1 month
  VAT was defined as the sum time of ventilator assisted post-surgery.
Days of ICU stay | 3 months
  Total number of days during ICU, reflecting overall recovery and the impact of any gastrointestinal or systemic complications.

CONTACTS AND LOCATIONS:
Overall Officials: Wenbo Meng, Principal Investigator — Hepatopancreatobiliary Surgery Institute of Gansu Province
Locations (1):
- Hepatopancreatobiliary Surgery Institute of Gansu Province, Lanzhou, Gansu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gallitto E, Sobocinski J, Mascoli C, Pini R, Fenelli C, Faggioli G, Haulon S, Gargiulo M. Fenestrated and Branched Thoraco-abdominal Endografting after Previous Open Abdominal Aortic Repair. Eur J Vasc Endovasc Surg. 2020 Dec;60(6):843-852. doi: 10.1016/j.ejvs.2020.07.071. Epub 2020 Aug 24. PMID 32855033
- [Background] Seilitz J, Edstrom M, Skoldberg M, Westerling-Andersson K, Kasim A, Renberg A, Jansson K, Friberg O, Axelsson B, Nilsson KF. Early Onset of Postoperative Gastrointestinal Dysfunction Is Associated With Unfavorable Outcome in Cardiac Surgery: A Prospective Observational Study. J Intensive Care Med. 2021 Nov;36(11):1264-1271. doi: 10.1177/0885066620946006. Epub 2020 Aug 10. PMID 32772778
- [Background] Reintam Blaser A, Malbrain ML, Starkopf J, Fruhwald S, Jakob SM, De Waele J, Braun JP, Poeze M, Spies C. Gastrointestinal function in intensive care patients: terminology, definitions and management. Recommendations of the ESICM Working Group on Abdominal Problems. Intensive Care Med. 2012 Mar;38(3):384-94. doi: 10.1007/s00134-011-2459-y. Epub 2012 Feb 7. PMID 22310869
- [Derived] Yang X, Lu N, Yang L, Li B, Zhou W, Li Y, Song B, Yuan J, Meng W. Impact of prolonged cardiopulmonary bypass on gastrointestinal complications in cardiac surgery: a retrospective cohort study. Perioper Med (Lond). 2025 Apr 15;14(1):42. doi: 10.1186/s13741-025-00524-w. PMID 40234981